CLINICAL TRIAL: NCT07317076
Title: Compression Anastomosis Using the GT Metabolic Magnet System in Adults With Gastrointestinal Disorders (GT Metabolic Magnet System Study)
Brief Title: GT Metabolic Magnet System in Adults With Gastrointestinal Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-020
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Gastric Outlet Obstruction; Small Bowel Obstruction; Superior Mesenteric Artery Syndrome
Keywords: Magnet System; GT Metabolic Solutions, Inc.
MeSH Terms: conditions — Gastric Outlet Obstruction; Superior Mesenteric Artery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnet System (Experimental): GT Metabolic Magnet System comprised of GT Metabolic Magnet System ("Magnet System")
  Interventions: Device: Magnet System

INTERVENTIONS:
Device: Magnet System — Magnetic compression anastomoses for intestinal diversion in subjects with small bowel obstruction, gastric outlet obstruction, or superior mesenteric artery syndrome.

SUMMARY:
Evaluate the performance and safety of the GT Metabolic Magnet System for the creation of side-to-side compression anastomosis in the stomach and/or small bowel in conditions requiring an anastomosis as part of the underlying clinical treatment.

DETAILED DESCRIPTION:
Evaluate the performance and safety of the Magnet System as a surgical tool for anastomosis in participants who have partial small bowel obstruction, SMAS, or GOO due to their similarities (they all involve a physical impediment (e.g., compression of the intestinal lumen) and/or mechanical blockage of the GI tract).

ELIGIBILITY:
Inclusion Criteria:

* Indicated for gastrointestinal surgery requiring a gastric and/or small bowel anastomosis, without need for immediate lumen patency, and meets one of the following criteria:

  1. Superior mesenteric artery syndrome (SMAS); OR
  2. Gastric outlet obstruction (GOO); OR
  3. Partial small bowel obstruction.
* Meets the surgical clearance requirements as governed by the investigator's institution.
* If a child-bearing female, subject must commit to not becoming pregnant and agree to use contraception for the duration of the study.

Exclusion Criteria:

* Other gastrointestinal or abdominal surgeries planned concurrently or within the study follow-up period (e.g., bariatric surgery such as sleeve gastrectomy).
* Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contraindicate the anastomosis or study procedure, including scarring and abnormal anatomy at the anastomosis sites.
* Any anomaly precluding gastrointestinal access by gastroscope / endoscope, catheters, and associated manipulation techniques for device placement.
* Any condition or disease that precludes laparoscopic surgery.
* Implantable pacemaker, defibrillator, other active and/or metallic implant that may interfere with or be adversely impacted by a temporary magnetic implant (Magnet System) and associated procedures.
* Unhealed ulcers, bleeding lesions, tumor, diseased tissue or any other lesion at or distal to the target Magnet deployment sites.
* Any need for immediate lumen patency while the anastomosis is formed.
* History of prior or current malignancy.
* Expected need for Magnetic Resonance Imaging (MRI) within the first 3 months post-procedure (or before if Magnet expulsion is confirmed radiologically).
* Known allergies to the device components (including the biofragmentable material PGLA or similar compounds) or contrast media.
* Pregnant, lactating, or planning pregnancy during the clinical investigation and follow up period.
* Currently participating in an investigational drug, biologic, or medical device or other interventional clinical study.
* Presence of other anatomic or comorbid conditions, or medical, social or psychological conditions that, in the investigator's opinion, could limit the participant's ability to participate in the clinical investigation or to comply with follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Magnet Placement | 1 day
  Placement and connection of two intraluminal Magnet.
Natural Magnet Passage | 90 days
  Successful passage of magnets without surgical reintervention
Anastomosis Patency | 90 days
  Creation of a patent anastomosis confirmed radiologically.

CONTACTS AND LOCATIONS:
Locations (1):
- Westmount Surgical Center, Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No